CLINICAL TRIAL: NCT04058171
Title: Validation of a Treadmill Walking Test to Discriminate Neurogenic Claudication From Vascular Claudication
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Principal investigator, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-2017-claudication
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Spinal Stenosis Lumbar; Low Back Pain; Peripheral Artery Disease; Claudication
Keywords: Walking capacity; Walking posture; Diagnostic test
MeSH Terms: conditions — Low Back Pain; Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LSS group: Participants with a diagnosis of lumbar spinal stenosis
  Interventions: Diagnostic Test: Treadmill walking test
- PAD group: Participants with a diagnosis of peripheral artery disease
  Interventions: Diagnostic Test: Treadmill walking test
- LBP group: Participants with a diagnosis of non specific low back pain
  Interventions: Diagnostic Test: Treadmill walking test

INTERVENTIONS:
Diagnostic Test: Treadmill walking test — Participants will be invited to walk on a treadmill at a speed of 1,2 mph for at most five minutes for both conditions (straight walking posture and inclined walking posture). Each walking posture condition will be followed by a rest time of five minutes in sitting position. Conditions were randomized in each group using a computer-generated sequence.

SUMMARY:
The first aim of this study was to elaborate and validate a treadmill walking test that would help discriminate between neurogenic claudication from vascular claudication. The second objective of this study is to determine if the treadmill walking test can discriminate spinal stenosis from low back pain with radiating pain in lower limb.

DETAILED DESCRIPTION:
To date, an important challenge that clinicians hare facing in the assessment and diagnosis of intermittent claudication is that pathologies associated with vascular or neurogenic claudication can coexist in the same patient. Differentiation between both origins can be difficult due to variable signs and symptoms which can be atypical.

The first aim of this study was to elaborate and validate a treadmill walking test that would help discriminate between neurogenic claudication from vascular claudication. The second objective of this study is to determine if the treadmill walking test can discriminate spinal stenosis from low back pain with radiating pain in lower limb. 60 participants (20 with spinal stenosis, 20 with peripheral artery disease and 20 with non-specific low back pain) will be recruited. Participants will be invited to walk on a treadmill at a speed of 1,2 mph for a maximum of five minutes for both tasks (straight walking posture and inclined walking posture). Each walking task will be followed by a rest time of five minutes in sitting position. It is hypothesized that walking time difference for the occurrence of pain and for pain relief will be sensitive and specific to pathologies and help to discriminate lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

Lumbar spinal stenosis (LSS) group :

* Central stenosis
* Pain in at least one leg
* Neurological signs in the lower limbs (numbness or tingling)
* Weaknesses in the lower limb
* Pain relieved by sitting or bending the trunk

Peripheral artery disease (PAD) group :

* Claudication while walking
* Ankle-brachial index < 0.9
* Pain relieved by rest

Low back pain (LBP) :

* Pain radiating in the lower limb
* Weaknesses
* Pain relieved by sitting

Exclusion Criteria:

* Foraminal stenosis
* Spinal stenosis with predominant back pain
* Symptomatic disc herniation
* Previous lumbar surgery
* Previous vascular surgery
* Type 1 diabetes
* Knee or hip osteoarthritis
* Hip or knee arthroplasty
* Inability to provide free and informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurogenic or vascular claudication
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Walking time | Time first back or leg pain (vary between participants from 0 secondes to 300 secondes and is determine by the occurence of leg or back pain), Through the walking test completion

SECONDARY OUTCOMES:
Leg and back Pain (Visual analog scale) | Before the walking test, through the walking test completion, at 2:30 minutes of rest, at 5 minutes of rest
  leg and back pain using a 0-10 points scale
Walking impairment Questionnaire (WIQ) | day 1, before the walking test (this is a transversal study)
  WIQdistance subscale score range from 0 to 100%, WIQspeed subscale score range from 0 to 100%, WIQstairs subscale score range from 0 to 100%, WIQ total score combining distance,speed and stairs subscale range from 0 to 100% Higher values indicate better outcome
Tampa Scale of kinesiophobia | day 1, before the walking test (this is a transversal study)
  Questionnaire, Total score range from 17 to 68, Higher score indicate a worst outcome
Quality of life of participants | day 1, before the walking test (this is a transversal study)
  EuroQol 5 dimension (EQ-5D), each section (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) has a score ranging from 1 to 3 and higher values indicate a worst outcome
Impact of pain, function and surgery satisfaction | day 1, before the walking test (this is a transversal study)
  French-Canadian adaptation of the Swiss Spinal Stenosis Questionnaire Pain subscale score range from 7 to 35 with higher values indicate a worst outcome, Function subscale score range from 5 to 20 with higher values indicate a worst outcome, Satisfaction subscale score range from 6 to 24 with higher values indicate a worst outcome. The total score is composed of the three subscales and range from 18 to 79.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houle M, O'Shaughnessy J, Tetreau C, Chatillon CE, Marchand AA, Descarreaux M. Comparison of walking variations during treadmill walking test between neurogenic and vascular claudication: a crossover study. Chiropr Man Therap. 2021 Jul 15;29(1):24. doi: 10.1186/s12998-021-00382-5. PMID 34266463